CLINICAL TRIAL: NCT03330951
Title: Glycemic Control and Iron Status in Diabetic Pregnancies - a Study of New Markers
Status: Completed | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: SUS-ID580
Record Dates: First submitted 2016-11-17; First posted 2017-11-06 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2018-12

CONDITIONS: Diabetes Mellitus Pregnancy
Keywords: HbA1c; Glycated albumin
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study at the Obstetrical outpatient clinic at Stavanger University Hospital. The main goal is to compare the current marker of glycemic control (glycated hemoglobin A1c, HbA1c) with glycated albumin in pregnancies with pregestational diabetes mellitus.

Women with diabetes are at increased risk for adverse pregnancy outcomes. With improved glycemic control, the risk decreases. Glycated albumin is suggested to be a better marker for monitoring glycemic control in pregnancies because it reflects blood glucose for a shorter period than HbA1c (3 versus 8-12 weeks). Other studies have shown that HbA1c increases in pregnancy because of iron deficiency. The investigators want to investigate HbA1c, glycated albumin and iron status in diabetic pregnancies. The investigators will compare HbA1c and glycated albumin throughout pregnancy with the patient's own blood glucose measurements or data from CGM (continuous blood glucose monitoring). Blood samples for HbA1c and glycated albumin will be taken 6 times during pregnancy (week 12, 20, 24, 28, 32, 36).

ELIGIBILITY:
Inclusion Criteria:

* pregestational diabetes mellitus
* singleton pregnancy
* follow-up at Stavanger University Hospital in pregnancy

Exclusion Criteria:

* gestational diabetes
* twin pregnancies

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women with pregestational diabetes mellitus
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Glycemic Control markers in pregnancy | throughout pregnancy, gestational week 12-36.
  Compare HbA1c and glycated albumin to blood sugar measurements

SECONDARY OUTCOMES:
Iron status in diabetic pregnancy, | throughout pregnancy, gestational week 12-36.
  Compare current markers of iron status with hepcidin throghout diabetic pregnancies by analyses of blood samples in gestational week 12, 20, 24, 28, 32 and 36.
Preterm delivery | at delivery.
  Register pregnancy outcomes. Delivery before gestational week 37 will be registered. Data will be collected from journals.
Preeclampsia | From gestational week 20 to 1 week after delivery.
  Register pregnancy outcomes. New onset systolic blood pressure >140, diastolic blood pressure >90 after gestational week 20 and proteinuria 2+ according to urine dipstick, will be registered as preeclampsia
Induction of labour | At delivery.
  Register pregnancy outcome. Induction of Labour and indication for induction will be registered.
APGAR | At delivery.
  Register pregnancy outcome. APGAR score (Appearance, Pulse, Grimace, Activity, Respiration) of the newborn will be registered for 1 minute, 5 minute and 10 minutes after delivery.
Birth weight | At delivery.
  Register pregnancy outcome. Birth weight (gram) of the newborn will be registered.
Admission to neonatal intensive care unit | At delivery.
  Register pregnancy outcome. Admission to neonatal intensive care unit will be registered.

CONTACTS AND LOCATIONS:
Overall Officials: Johanne Toft, MD, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Rogaland, Norway

IPD SHARING:
Plan to Share IPD: No